CLINICAL TRIAL: NCT02592460
Title: Impact on Pain of a Preoperative Polyamines-poor Diet After Orthopedic Surgery of the Foot
Brief Title: Postoperative Pain and Polyamines-poor Diet (DOLAMINE)
Acronym: DOLAMINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WGF_2014-2
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2017-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- poor-polyamines diet (Experimental)
  Interventions: Other: poor-polyamines diet
- high-polyamines diet (Active Comparator)
  Interventions: Other: high polyamines diet

INTERVENTIONS:
Other: poor-polyamines diet — Patients in this will receive a poor-polyamines diet during a week before and a week after foot surgery
  Arms: poor-polyamines diet
Other: high polyamines diet — Patients in this will receive a high-polyamines diet during a week before and a week after foot surgery
  Arms: high-polyamines diet

SUMMARY:
Animal studies have shown that the level of pain sensitivity is highly dependent on the amount of polyamines in food. This fundamental observation of a nutritional approach to pain led the authors to develop diets completely depleted in polyamines whose anti-nociceptive properties have been confirmed in animals.

Postoperative pain after foot surgery are currently fairly well controlled but at the cost of a high consumption of grade II analgesics which is associated with a high rate of side effects (nausea, vomiting ...). The investigators' hypothesis is that a diet low in polyamines may have an additive effect on pain control and reduce the consumption of level 2 analgesics.

The objective of this study is to show the efficacy of a polyamines-poor diet on postoperative pain in ambulatory surgery of the foot.

ELIGIBILITY:
Inclusion Criteria:

* foot ambulatory orthopedic surgery
* surgery scheduled at least 10 days after the inclusion consultation

Exclusion Criteria:

* other diet susceptible to interfere with the poor or high-polyamines diets (e.g. diabetic patients)
* contraindication to tramadol or to NSAIDs
* pregnant or breastfeeding woman
* patient under legal protection
* patient's opposition to participate in the study
* poor understanding of French
* absence of affiliation to social security
* participation to another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients whose worst pain, as measured on an visual analogic scale ranging from 0 mm to 100 mm, was at least once rated as 30 mm or more. | Eight days after surgery
  The worst pain will be assessed retrospectively the eighth day after surgery

SECONDARY OUTCOMES:
Percentage of patients with a need for grade II analgesics | Eighth day after surgery
Overall tramadol consumption , expressed in mg. | Eight days after surgery
Worst pain, expressed in mm, measured on an visual analogic scale ranging from 0 mm to 100 mm | Eight days after surgery
  The worst pain will be assessed retrospectively the eighth day after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe hospitalier Diaconesses Croix Saint Simon, Paris, Île-de-France Region, France